CLINICAL TRIAL: NCT02209428
Title: A Prospective Cohort to Study the Effect of Postoperative Upfront Temozolomide Chemotherapy on IDH Mutational Low Grade Gliomas in Eloquent Areas
Brief Title: A Prospective Cohort to Study the Effect of Temozolomide on IDH Mutational Low Grade Gliomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jinsong Wu, Professor, Huashan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY2014-182
Record Dates: First submitted 2014-07-30; First posted 2014-08-05 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Astrocytoma; Oligodendroglioma; Oligoastrocytoma
Keywords: Temozolomide; IDH mutation; Low grade glioma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma | interventions — Temozolomide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IDH wild type (Active Comparator): Patients with IDH wild type, according to the result of genetic sequencing of their surgical resected specimens. Intervention: oral temozolomide, 75 mg/m2/day for 21 days repeated every 4 weeks, 6 cycles.
  Interventions: Drug: Temozolomide
- IDH mutation (Experimental): Patients with IDH mutations, according to the result of genetic sequencing of their surgical resected specimens. Intervention: oral temozolomide, 75 mg/m2/day for 21 days repeated every 4 weeks, 6 cycles.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — 75 mg/m2/day for 21 days repeated every 4 weeks, 6 cycles.
  Other Names: Temodar; Temodal

SUMMARY:
Low grade gliomas (LGGs) are the most common primary central nervous system malignancies. Brain surgeries with the most possible extent of resection are endeavored to achieve longer survivals in LGG patients. For patients with tumor located in eloquent areas so that gross total resection is not applicable, National Comprehensive Cancer Network (NCCN) 2013 guidelines assigned both radiotherapy or chemotherapy as adjuvant treatments of low grade glioma following surgeries. Retrospective studies have suggested that temozolomide (an oral chemotherapeutics) chemotherapy have good effects on the control of tumor progression or recurrence in LGG patients after surgeries, especially in those with isocitrate dehydrogenase (IDH) gene mutations.

Therefore, our prospective cohort study is to provide a higher level(IIb) of evidence for the correlation between IDH mutation and the responsiveness to up-front adjuvant metronomic temozolomide chemotherapy in young patients with LGG located in eloquent brain areas. And hopefully justify future RCTs with comparison between effects of adjuvant radiotherapy and chemotherapy in these patients.

DETAILED DESCRIPTION:
Low grade gliomas, according to the 2007 WHO classification of tumors of the central nervous system, include astrocytomas, oligodendrogliomas, and oligoastrocytomas. It contributes to 25% of diffuse gliomas and 15% of all gliomas in adults. The majority of age group that is the most vulnerable to this neoplasm is from 30-45 years old. Median survival is usually 5-12 years, but can be prolonged up to 20 years under optimal treatment strategies. National Comprehensive Cancer Network (NCCN) and Chinese Guideline for Gliomas 2012 both point out that for LGG patients in low-risk group (oligodendrogliomas or oligoastrocytomas; no more than 40 years old; KPS 80 and higher; tumor size less than 6cm; no or minor neurological deficits), "wait and see" strategy could be considered after gross total resection; but when the tumors are in eloquent areas so that gross total resections are not applicable, the standard strategies for this specific group of patients are maximum safely resection with adjuvant treatments (radiotherapy and/or chemotherapy). Conventionally, radiotherapy is used as adjuvant treatment after surgeries. However, a recent phase III randomized trial comparing early versus later irradiation has demonstrated that early adjuvant radiotherapy had no significant impact on overall survival. Moreover, radiotherapy brings as much side effects as its control of tumor recurrence. It inevitably jeopardizes patients, especially young ones, with post-radiation cognitive deficits, which impair their social functions. On the other hand, chemotherapy could be a safer adjuvant treatment for LGG. Several phase II and III studies demonstrated that single chemotherapy is effective for treating LGG, with 50-75% response rate (including minor response), and 24-48 months of median duration of response.PCV regimen (procarbazine-CCNU-vincristine), which is administrated intravenously, used to be considered standard for LGG (oligodendrogliomas and oligoastrocytomas) chemotherapy, but now temozolomide (TMZ), an oral alkylating agent, with relatively less side effects than PCV regimen, is gaining gradual acceptance. Now we propose up-front adjuvant chemotherapy to achieve the effect of early tumor control as well as avoidance or postponement of adverse effects caused by premature adjuvant radiotherapy.

As for different schedules of temozolomide, a systematic review suggested an indication that metronomic regimens of TMZ (75 mg/m2/day for 21 days repeated every 4 weeks) result in better PFS and response rate when compared to the conventional standard 5 day regimen (200 mg/m2/day for 5 days, repeated every 4 weeks), despite of insufficient available data and study heterogeneity, thus justifying future well designed trials to verify the efficacy of the metronomic regimen. More frequent administration of TMZ will lead to MGMT (O6-methylguanine DNA methyl transferase) depletion and render higher levels of O6-methylated DNA adducts, thus reducing the chemotherapeutic resistance.

The spontaneous behavior of LGGs, as well as their response to therapy, is difficult to predict, and their outcome is highly variable. These clinical features are closely relevant to their genetic characteristics, including IDH (isocitrate dehydrogenase) gene, with 2 subtypes, IDH1 and IDH2 (less common). These genetic mutations occur in more than 70% primary LGGs. And its prognostic significance of gliomas has been reported in the New England Journal of Medicine, Journal of Clinical Oncology, and Neuro-oncology. A retrospective study suggested its predictive value of high LGGs sensitivity to TMZ. Basic research provided us the rationale that overexpression of wild IDH1 gene resulted in chemotherapy resistance to a high dose of TMZ in vivo and in vitro, while IDH1 mutation caused cell cycle arrest in G1 stage, with a compromised ability of proliferation and invasion, raising sensitivity to chemotherapy.

During our previous clinical practice, it is interesting to reveal the consistence of IDH mutation, MGMT methylation and 1p19q co-deletion in WHO Grade II and Grade III gliomas. It theoretically acknowledged potential higher sensitivity of TMZ chemotherapy in LGGs.

In order to verify the predictive significance of IDH mutation for a higher sensitivity of LGGs in eloquent areas which entail gross total resection inapplicable, higher level of evidence should be provided. And recent RANO (response assessment in neuro-oncology) revised guidelines for evaluations of objective response rate, cognitive functions, and quality of life have better facilitated standard trials.

ELIGIBILITY:
Inclusion Criteria:

* 18 years < age ≤ 40 years, both genders.
* No neurologic cognitive deficits (MMSE ≥ 27), no psychiatric abnormalities before surgery, pre-operative KPS ≥ 80.
* Tumors located in eloquent areas or deeply located nuclei, rendering radiological complete resection inapplicable, according to updated standards of extent of resection: as for non-enhancing LGG, postoperative MRI within 72h shows absence of any preoperative T2/FLAIR signal changes - complete resection; and for enhancing LGG, postoperative MRI shows total removal of preoperative enhancing tissue - complete resection of enhancing tumor; and total removal of enhancing and non-enhancing tissues (T2/FLAIR) - complete resection of detectable tumor.
* Post-operative histological pathology confirms LGGs (astrocytomas, oligodendrogliomas, or oligoastrocytomas, 2007 WHO classification Grade II).
* No contraindications to TMZ chemotherapy.
* Informed consent to TMZ chemotherapy.

Exclusion Criteria:

* Tumor involves more than 3 cerebral lobes (gliomatosis or multiple gliomas).
* Tumor is complicated with other intracranial neoplasms (e.g. metastatic tumors or meningiomas).
* Tumor is complicated with systematic malignancies.
* Dysfunctions of other vital organs: liver and kidney (ALT﹥40U/L, AST > 40U/L, creatinine > 97-106μmol/L, urea nitrogen > 7.1mmol/L, or other lab abnormalities); Heart (NYHA II-IV); Lungs (hypoxemia).
* Physiological pregnancy.
* Participate in other clinical trials at meantime.
* History of severe anaphylaxis.
* Voluntarily quit or decline chemotherapy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2014-06; Primary Completion 2019-04 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate, ORR | Within 72 hours after surgery, at the beginning of chemotherapy, every 2 months thereafter up to a year, every 3-6 months after a year, until the first documented progression or date of death from any cause, whichever came first, up to 2 years.
  According to the revised RANO criteria (M J van den Bent, et al. 2011), compared to residual tumor volume calculated with iMRI T2/Flair right after surgery and before up-front adjuvant chemotherapy (Baseline tumor volume):
  Complete response (CR): disappearance of abnormality Partial response (PR): no less than 50% reduction Minimal response (MR): no less than 25% but less than 50% reduction Stable disease (SD): less than 25% reduction also less than 25% increase Progressive disease (PD): no less than 25% increase
  Enhanced T1-weighted imaging, magnetic resonance spectroscopy (MRS), Diffusion tensor imaging (DTI) and perfusion-weighted imaging (PWI) will also be utilized to detect progressions.
Velocity of Diameter Evolution, VDE | Within 72 hours after surgery, at the beginning of chemotherapy, every 2 months thereafter up to a year, every 3-6 months after a year, until the first documented progression or date of death from any cause, whichever came first, up to 2 years.
  According to the Definition of New Endpoints by E. Mandonnet et al, 2013, VDE is calculated with formula D = (2 × V)^1/3, (V= tumor volume).
  Uncontrolled: unchanged or increased VDE compared to baseline VDE. Slowed down: decreased VDE compared to baseline VDE, but still positive. Stabilized: VDE is close to 0 mm/year. Reversed: negative VDE. Treatment escape and relapse: re-growth of the tumor greater than 2 mm, during the course of chemotherapy and after the end of chemotherapy, respectively.
  Intensity of response (IOR): how much the diameter has been reduced by the therapy.
  Duration of response (DOR): the time period between treatment onset and treatment escape or relapse. If Replapse (25% increase/VDE>2mm/Maligmant enhancement), start 2° treatment: Second surgery or radiotherapy or salvage chemotherapy

SECONDARY OUTCOMES:
Progression free survival (PFS)-6, -12, -24 | 6, 12 and 24 months after the 1st cycle of chemotherapy
  The survival rate of followed patients without progressive disease (PD) 6, 12, and 24 months after the 1st cycle of chemotherapy
Cognitive functions | At the beginning of chemotherapy, every 2 months thereafter up to a year, and every 3-6 months after a year of follow-up, until the first documented (malignant) progression or date of death from any cause, whichever came first, up to 2 years.
  Test battery:
  Measured with Minimal Mental State Examination (MMSE); Hopkins verbal learning test-revised; Trail making test, part A and B; Multilingual aphasia examination controlled oral word association
Quality of life (QoL) | At the beginnning of chemotherapy, every 2 months thereafter up to a year, and every 3-6 months after a year of follow-up, until the first documented (malignant) progression or date of death from any cause, whichever came first, up to 2 years.
  Measured with EORTC QLQ-C30 and EORTC-BN20. Duration of response with good quality of life is defined as Time with good quality of life (TQL).
Adverse effect of chemotherapy | At the beginning of chemotherapy, every 2 months thereafter up to a year, until the first documented (malignant) progression or date of death from any cause, whichever came first, up to 2 years.
  Blood routine and kidney/liver functions
Malignant progression-free survival (MPFS) -6, -12, -24 | 6, 12 and 24 months after the 1st cycle of chemotherapy
  The survival rate of followed patients without any MRI T1 enhancing signals in 6, 12, and 24 months after the 1st cycle of chemotherapy
Symptom Burden | At the beginning of the chemotherapy, every 2 months thereafter up to a year, then every 3 months up to 2 years
  Measured with M.D. Anderson Symptom Inventory Brain Tumor Module, MDASI-BT.
Seizure activity | At the beginning of the chemotherapy, every 2 months thereafter up to a year, then every 3 months up to 2 years
  Measured by one neurologist, number and type of seizure and medication in the past month before each follow-up visit are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Wu, Professor, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Louis DN, Ohgaki H, Wiestler OD, Cavenee WK, Burger PC, Jouvet A, Scheithauer BW, Kleihues P. The 2007 WHO classification of tumours of the central nervous system. Acta Neuropathol. 2007 Aug;114(2):97-109. doi: 10.1007/s00401-007-0243-4. Epub 2007 Jul 6. PMID 17618441
- [Background] Viaccoz A, Lekoubou A, Ducray F. Chemotherapy in low-grade gliomas. Curr Opin Oncol. 2012 Nov;24(6):694-701. doi: 10.1097/CCO.0b013e328357f503. PMID 22913972
- [Background] Houillier C, Wang X, Kaloshi G, Mokhtari K, Guillevin R, Laffaire J, Paris S, Boisselier B, Idbaih A, Laigle-Donadey F, Hoang-Xuan K, Sanson M, Delattre JY. IDH1 or IDH2 mutations predict longer survival and response to temozolomide in low-grade gliomas. Neurology. 2010 Oct 26;75(17):1560-6. doi: 10.1212/WNL.0b013e3181f96282. PMID 20975057
- [Background] Vogelbaum MA, Jost S, Aghi MK, Heimberger AB, Sampson JH, Wen PY, Macdonald DR, Van den Bent MJ, Chang SM. Application of novel response/progression measures for surgically delivered therapies for gliomas: Response Assessment in Neuro-Oncology (RANO) Working Group. Neurosurgery. 2012 Jan;70(1):234-43; discussion 243-4. doi: 10.1227/NEU.0b013e318223f5a7. PMID 21593697
- [Background] Wang JB, Dong DF, Wang MD, Gao K. IDH1 overexpression induced chemotherapy resistance and IDH1 mutation enhanced chemotherapy sensitivity in Glioma cells in vitro and in vivo. Asian Pac J Cancer Prev. 2014;15(1):427-32. doi: 10.7314/apjcp.2014.15.1.427. PMID 24528069
- [Background] Nabors LB, Portnow J, Ahluwalia M, Baehring J, Brem H, Brem S, Butowski N, Campian JL, Clark SW, Fabiano AJ, Forsyth P, Hattangadi-Gluth J, Holdhoff M, Horbinski C, Junck L, Kaley T, Kumthekar P, Loeffler JS, Mrugala MM, Nagpal S, Pandey M, Parney I, Peters K, Puduvalli VK, Robins I, Rockhill J, Rusthoven C, Shonka N, Shrieve DC, Swinnen LJ, Weiss S, Wen PY, Willmarth NE, Bergman MA, Darlow SD. Central Nervous System Cancers, Version 3.2020, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2020 Nov 2;18(11):1537-1570. doi: 10.6004/jnccn.2020.0052. PMID 33152694
- [Background] van den Bent MJ, Taphoorn MJ, Brandes AA, Menten J, Stupp R, Frenay M, Chinot O, Kros JM, van der Rijt CC, Vecht ChJ, Allgeier A, Gorlia T; European Organization for Research and Treatment of Cancer Brain Tumor Group. Phase II study of first-line chemotherapy with temozolomide in recurrent oligodendroglial tumors: the European Organization for Research and Treatment of Cancer Brain Tumor Group Study 26971. J Clin Oncol. 2003 Jul 1;21(13):2525-8. doi: 10.1200/JCO.2003.12.015. PMID 12829671
- [Background] Brada M, Viviers L, Abson C, Hines F, Britton J, Ashley S, Sardell S, Traish D, Gonsalves A, Wilkins P, Westbury C. Phase II study of primary temozolomide chemotherapy in patients with WHO grade II gliomas. Ann Oncol. 2003 Dec;14(12):1715-21. doi: 10.1093/annonc/mdg371. PMID 14630674
- [Background] Lashkari HP, Saso S, Moreno L, Athanasiou T, Zacharoulis S. Using different schedules of Temozolomide to treat low grade gliomas: systematic review of their efficacy and toxicity. J Neurooncol. 2011 Nov;105(2):135-47. doi: 10.1007/s11060-011-0657-7. Epub 2011 Jul 5. PMID 21748491
- [Background] Yan H, Parsons DW, Jin G, McLendon R, Rasheed BA, Yuan W, Kos I, Batinic-Haberle I, Jones S, Riggins GJ, Friedman H, Friedman A, Reardon D, Herndon J, Kinzler KW, Velculescu VE, Vogelstein B, Bigner DD. IDH1 and IDH2 mutations in gliomas. N Engl J Med. 2009 Feb 19;360(8):765-73. doi: 10.1056/NEJMoa0808710. PMID 19228619
- [Background] Sanson M, Marie Y, Paris S, Idbaih A, Laffaire J, Ducray F, El Hallani S, Boisselier B, Mokhtari K, Hoang-Xuan K, Delattre JY. Isocitrate dehydrogenase 1 codon 132 mutation is an important prognostic biomarker in gliomas. J Clin Oncol. 2009 Sep 1;27(25):4150-4. doi: 10.1200/JCO.2009.21.9832. Epub 2009 Jul 27. PMID 19636000
- [Background] Ichimura K, Pearson DM, Kocialkowski S, Backlund LM, Chan R, Jones DT, Collins VP. IDH1 mutations are present in the majority of common adult gliomas but rare in primary glioblastomas. Neuro Oncol. 2009 Aug;11(4):341-7. doi: 10.1215/15228517-2009-025. Epub 2009 May 12. PMID 19435942
- [Background] van den Bent MJ, Wefel JS, Schiff D, Taphoorn MJ, Jaeckle K, Junck L, Armstrong T, Choucair A, Waldman AD, Gorlia T, Chamberlain M, Baumert BG, Vogelbaum MA, Macdonald DR, Reardon DA, Wen PY, Chang SM, Jacobs AH. Response assessment in neuro-oncology (a report of the RANO group): assessment of outcome in trials of diffuse low-grade gliomas. Lancet Oncol. 2011 Jun;12(6):583-93. doi: 10.1016/S1470-2045(11)70057-2. Epub 2011 Apr 5. PMID 21474379
- [Background] E. Mandonnet et al. Toward the Definition of New Endpoints. H. Duffau (ed.), Diffuse Low-Grade Gliomas in Adults, DOI 10.1007/978-1-4471-2213-5_29, Springer-Verlag London 2013
- [Background] Aibaidula A, Lu JF, Wu JS, Zou HJ, Chen H, Wang YQ, Qin ZY, Yao Y, Gong Y, Che XM, Zhong P, Li SQ, Bao WM, Mao Y, Zhou LF. Establishment and maintenance of a standardized glioma tissue bank: Huashan experience. Cell Tissue Bank. 2015 Jun;16(2):271-81. doi: 10.1007/s10561-014-9459-4. Epub 2014 Jun 15. PMID 24929994
- [Background] van den Bent MJ, Afra D, de Witte O, Ben Hassel M, Schraub S, Hoang-Xuan K, Malmstrom PO, Collette L, Pierart M, Mirimanoff R, Karim AB; EORTC Radiotherapy and Brain Tumor Groups and the UK Medical Research Council. Long-term efficacy of early versus delayed radiotherapy for low-grade astrocytoma and oligodendroglioma in adults: the EORTC 22845 randomised trial. Lancet. 2005 Sep 17-23;366(9490):985-90. doi: 10.1016/S0140-6736(05)67070-5. PMID 16168780